CLINICAL TRIAL: NCT07320495
Title: Efficacy and Safety of the APGO Algorithm for Automated Insulin Delivery: The RENEW Study
Brief Title: Efficacy and Safety of the APGO Algorithm for Automated Insulin Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RENEW
Record Dates: First submitted 2025-12-03; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus Type 1
Keywords: automated insulin delivery system; patch pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Patients with TouchCare Nano A8 insulin pump with the APGO system (Experimental): Patients with type 1 diabetes, who initiated use of the TouchCare Nano A8 insulin pump with the APGO system.
  Interventions: Device: Device: Insulin pump TouchCare Nano A8 with the APGO system

INTERVENTIONS:
Device: Device: Insulin pump TouchCare Nano A8 with the APGO system — Insulin pump Medtrum TouchCare Nano A8 with the APGO algorithm is the only patch pump-based automated insulin delivery system available in the Czech Republic.

SUMMARY:
The Medtrum TouchCare Nano system with the APGO algorithm is the only patch pump-based automated insulin delivery system available in the Czech Republic. However, until now, no prospective clinical study has evaluated its efficacy and safety under real-world conditions. The RENEW study is the first to address this topic.

ELIGIBILITY:
Inclusion Criteria:

* patients with T1D
* type 1 diabetes for ≥1 years
* ≥ 18 years old
* written informed consent prior to starting study related activity

Exclusion Criteria:

* severe noncompliance
* lactation, pregnancy, intending to become pregnant during study
* use of medication with effects on carbohydrate metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2027-06-19 (Estimated); Study Completion 2028-06-19 (Estimated)

PRIMARY OUTCOMES:
Changes in glycated haemoglobin (HbA1c) | Up to 24 months
  Differences between HbA1c values in the Visit 0 and Visit 24
Changes in percentage of time in target ranges 3,9-10,0 mmol/L (70-180 mg/dl) | Up to 24 months
  Differences between percentage of time in target ranges in the Visit 0 and Visit 24

SECONDARY OUTCOMES:
Changes in percentage of time in hypoglycemic ranges <3.9 mmol/L (70 mg/dl) and <3.0 mmol/L (54 mg/dl) | Up to 24 months
  Differences between percentage of time in hypoglycemic ranges in the Visit 0 and Visit 24
Changes in percentage of time in hyperglycemic ranges >10,0 mmol/L (180 mg/dl) and >13,9 mmol/L (250 mg/dl) | Up to 24 months
  Differences between percentage of time in hyperglycemic ranges in the Visit 0 and Visit 24
Changes in percentage of time in tight target ranges 3,9-7,8 mmol/L (70-140 mg/dl) | Up to 24 months
  Differences between percentage of time in tight target ranges in the Visit 0 and Visit 24
Changes in average glycemia (mmol/L) | Up to 24 months
  Differences between average glycemia in the Visit 0 and Visit 24
Changes in estimated glycated haemoglobin GMI (%) | Up to 24 months
  Differences between estimated glycated haemoglobin GMI in the Visit 0 and Visit 24
Changes in glycemic variability expressed as the coefficient of variation (%) | Up to 24 months
  Differences between glycemic variability in the Visit 0 and Visit 24
Time spent in automated insulin delivery mode | Up to 24 months
  Expressed as percentage of time

CONTACTS AND LOCATIONS:
Locations (1):
- 3rd Department of Internal Medicine, 1st Faculty of Medicine, Charles University, Prague, Czechia, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rimon MTI, Hasan MW, Hassan MF, Cesmeci S. Advancements in Insulin Pumps: A Comprehensive Exploration of Insulin Pump Systems, Technologies, and Future Directions. Pharmaceutics. 2024 Jul 15;16(7):944. doi: 10.3390/pharmaceutics16070944. PMID 39065641
- [Result] Ginsberg BH. Patch Pumps for Insulin. J Diabetes Sci Technol. 2019 Jan;13(1):27-33. doi: 10.1177/1932296818786513. Epub 2018 Aug 2. PMID 30070604
- [Result] Kulzer B, Freckmann G, Heinemann L, Schnell O, Hinzmann R, Ziegler R. Patch Pumps: What are the advantages for people with diabetes? Diabetes Res Clin Pract. 2022 May;187:109858. doi: 10.1016/j.diabres.2022.109858. Epub 2022 Apr 1. PMID 35367523